CLINICAL TRIAL: NCT04695587
Title: The Role of Sympathetic Tone Regarding the Anatomical and Functional Recovery of the Left Ventricle in TakoTsubo Syndrome
Acronym: SYMPATAK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Collaborators: Naval Hospital, Athens (Other); General Hospital of Athens Elpis (Other); 401 General Military Hospital of Athens (Other); 251 Hellenic Air Force & VA General Hospital (Other); Evangelismos Hospital (Other); Alexandra Hospital, Athens, Greece (Other); Sismanoglio General Hospital (Other); G.Gennimatas General Hospital (Other); Laikο General Hospital, Athens (Other); Tzaneio General Hospital (Other); Thriasio General Hospital of Elefsina (Other); National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Tsioufis, Professor in Cardiology, Hippocration General Hospital
Other Study IDs: 1920004531
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Takotsubo Cardiomyopathy
Keywords: sympathetic tone; autonomic nervous system; takotsubo; stress cardiomyopathy; 123MIBG; MSNA; Heart Rate Variability; Blood Pressure Variability
MeSH Terms: conditions — Takotsubo Cardiomyopathy | interventions — Electrocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma biomarkers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TakoTsubo: Patients hospitalized with TakoTsubo syndrome according to the INTERTAK criteria
  Interventions: Diagnostic Test: 123 MIBG scintigraphy testing; Diagnostic Test: MSNA; Diagnostic Test: ABPM; Diagnostic Test: ECHO; Diagnostic Test: 24hour ECG; Diagnostic Test: CMR

INTERVENTIONS:
Diagnostic Test: 123 MIBG scintigraphy testing — 123 MIBG scintigraphy testing in subacute phase and 12 months after the acute episode in a subgroup of patients according to individualized needs.
Diagnostic Test: MSNA — MSNA in subacute phase and 12 months after the acute episode
Diagnostic Test: ABPM — ABPM in subacute phase and 12 months after the acute episode
Diagnostic Test: ECHO — ECHO in subacute phase and 12 months after the acute episode
Diagnostic Test: 24hour ECG — 24hour ECG in subacute phase and 12 months after the acute episode
Diagnostic Test: CMR — CMR in 12 months after the acute episode

SUMMARY:
TakoTsubo Syndrome (TTS) constitutes an increasingly recognised, heterogenous clinical entity which is associated with considerable short-term mortality. In addition, emerging evidence suggests that, in the long term, TTS can induce the expression of a phenotype similar to HFpEF . Apart from the typical (apical left ventricular) type, the current TTS definition has been expanded to also include the mid-ventricular, the basal and the focal type. Several previous studies on the typical form of the syndrome demonstrated that the principal underlying pathophysiology is sympathetic overactivation.

Purpose The aim of this study is to investigate the potential association between the sympathetic tone and the acute phase clinical features of TTS. Furthermore, the investigators aim at exploring possible correlations between the sympathetic tone activity and the diastolic dysfunction, a reported complication occurring one year after the acute phase.

This is a prospective observational study enrolling patients aged 18-85 years who fulfill the InterTaK diagnostic criteria and whose CMR within 14 days of the onset is not suggestive of an alternative diagnosis. All patients will be treated on individual basis according to the recent expert consensus statement for TTS. During the baseline evaluation the sympathetic tone will be assessed by means of Muscle Sympathetic Nerve Activity study (MSNA), heart rate and blood pressure variability parameters. Additionally, in a subgroup of participants sympathetic activity and cardiac sympathetic enervation will be evaluated with radioactive Iodine Metaiodobenzylguanidine scintigraphy (mIBG). Sequential echocardiography and CMR indices will be used for heart function and geometry assessment. The investigators will investigate the correlation between the sympathetic tone and the severity of cardiac dysfunction (systolic and diastolic) during the acute phase. Furthermore, the investigators will examine differences of the sympathetic tone effect in association with the localisation of the wall motion abnormality. Stress levels and quality of life will be assessed with respective validated questionnaires. The participants will be followed-up with quarterly clinic reviews for 12 months after the acute event. Baseline measurements will be repeated at the end of the follow-up period. Ethics approval has been obtained from the hospital ethical committee board.

The study results are expected to determine the role of the sympathetic tone on the extend, the severity and the localisation of cardiac dysfunction during the acute phase. They are also expected to demonstrate the role of the sympathetic tone on the long-lasting disorder that persists for months following the acute event.

DETAILED DESCRIPTION:
TakoTsubo syndrome is the acute cardiac disorder which mimics an acute coronary syndrome and presents with signs of acute heart failure. It refers to a reversible regional dysfunction of the left ventricular contractility which cannot be attributed to coronary artery disease. Cardiac magnetic resonance is generally recommended as superior to echocardiography as the method to differentiate subjects with myocarditis or subendocardial infarction, but also to detect limited areas of reduced contractility and intracardiac thrombi. Usually, the condition follows an intense stressful event (physical condition or emotional distress). The affected area is usually regional, however cases of focal or global dysfunction of the left ventricle as well as others with right heart involvement have been also described. To date, many potential pathophysiologic processes have been suggested. These are the epicardial spasm, the self-limited acute myocardial infarction, the coronary microcirculatory dysfunction, the left ventricular outflow obstruction and the direct toxicity of the circulating catecholamines. Despite the comprehensive study of this entity during the last three decades, none of the aforementioned mechanisms has been adequately validated. On the other hand, there is increasing evidence regarding the leading role of the sympathetic tone as a main contributor. This has been shown in studies with 123mIBG which demonstrate that during the subacute phase of the syndrome the regional sympathetic enervation appears to be dysfunctional and improves after the recovery of the left ventricular systolic function. On the contrary, the sympathetic tone appears to be increased during the acute phase. There are no data available regarding the sympathetic innervation later than the period of three months from the episode. The MSNA, despite being a useful method to evaluate the sympathetic tone, has been used in TakoTsubo syndrome published series only twice. The available results are conflicting as there was a group of patients whose estimated sympathetic tone, being evaluated with MSNA appeared to be lower during the subacute phase compared with the follow - up period after the systolic recovery of the left ventricle.

Some years ago, despite its initial severity on presentation, the syndrome was regarded as having a benign course. New data, support that Takotsubo syndrome is accompanied by significant morbidity and mortality. Its incidence is estimated at around 2% of the acute coronary syndromes. It is exceptionally high in post-menopausal women. The available data support that short-term mortality ranges around 4-6% and is comparable to the one of the acute coronary syndromes. The disappointing short-term prognosis reflects the increased epidemiological data of in-hospital morbidity.

According to the International Takotsubo Registry, the men to women ratio is 9:1. The two genders share similar clinical and demographic characteristics, however in men, the stressful preceded event is more often physical but in women emotional. Typically, Takotsubo patients compared with others suffering from acute coronary syndromes suffer more frequently from depression and anxious disorder. Of great interest are the results which refer to the long-term morbidity. In detail, there are data for patients one year after the episode of Takotsubo syndrome who despite the left ventricular systolic recovery, express symptoms, functional status and laboratory results compatible with cardiac dysfunction. These findings are accompanied by increased myocardial fibrosis measured in CMR studies and abnormal metabolic function shown in cardiac magnetic spectroscopy. Moreover, it is suggested that the remaining diastolic dysfunction predisposes to worse outcomes. In general, Takotsubo syndrome is exceptionally heterogenous in terms of clinical expression and outcomes.

Aim of this study The main target of this study is to evaluate the sympathetic tone in patients with Takotsubo syndrome and particularly its potential prognostic value regarding its clinical severity on admission but also the left ventricular remodeling (structural and functional) one year after the event. It will be the first registry held in Greece and will try to re-evaluate the value of MSNA as a way to estimate the sympathetic tone in this population. Moreover, the sympathetic tone and sympathetic innervation integrity will be evaluated in patients with other than the typical - apical form of the syndrome according to the recent classification.

Methods This is a prospective, non-interventional observational study which will enroll patients 18-85-year-old, who fulfil the InterTAK diagnostic criteria. The diagnosis will be confirmed with CMR and ECHO which will show the LV systolic recovery. The sympathetic tone will be assessed with heart rate and blood pressure variability, MSNA and 123mIBG. Baseline measurements will be done during a 14-day interval from the acute onset. These will be repeated one year after the event. Signed consent form will be obtained and cases that the symptoms were attributed to myocarditis or subendocardial infarction (CMR result) will be excluded. Patients with severe chronic kidney disease (eGFR < 30 ml/min), severe valvular disease, contraindication to perform any of the aforementioned measurements, chronic atrial fibrillation, permanent pacing, autonomic failure, pregnant or breastfeeding women, psychiatric disease which does not allow adequate co-operation or patients with life expectancy less than a year will not be enrolled. The enrolled cases will be followed up for one year. Data will be collected in a specific form (CRF). These include demographic and somatometric data, past medical history, hemodynamics and sympathetic tone measurements. In detail, the following parameters will be measured. Gender, height, body weight, waist - hip and neck circumference, stress levels (validated questionnaire), tobacco exposure, history of hypertension, diabetes, dyslipidemia, family history of cardiovascular disease. Additionally, the investigators will collect information about the concomitant coronary artery disease, heart failure, paroxysmal atrial fibrillation, chronic kidney disease, peripheral artery disease, sleep apnea, stroke. Moreover, vital signs on admission, ECG findings, ECHO results on admission, cath lab results and laboratory results (estimated renal function, lipids, serum glucose levels, uric acid levels, liver function tests, thyroid function tests, myocardial ischemia biomarkers, natriuretic peptids and inflammatory markers).

Sympathetic tone estimation:

Α. MSNA. After patient's stabilization the test will be performed and the derived data will be the number of bursts per min and the average bursts per 100 beats. The test will be repeated one year after the acute event.

B. 123 MIBG. Lugol solution will be administered prior to the scan for thyroid protection. After the MIBG administration planar view will be obtained at 15-20 min and this will be repeated 4 hours later together with tomographic scan with γ camera. The measured parameters will be the early and late heart to mediastinum ratio and the washout ratio.

C. ambulatory heart rate and blood pressure monitoring. Heart rate variability will be analyzed via Kubios software for linear parametric characterization of short-term and long-term heart rate variability. Blood pressure short-term variability will be expressed as SD, wSD, ARV, CV, tame rate of BP variation.

The left ventricle geometry and function will be assessed with:

A. CMR (pre enrollment and one year after the episode). LV, RV: ESV, EDV, RWMA, atrial volumes, tissue tracking: GLS, RS. T2W-Triple IR/STIR, early and late gadolinium enhancement.

B. ECHO (acute phase of Takotsubo syndrome, one year after the event). LVEF, E, A, E', A', LA vol, GLS

For data analysis, SPSS 24.0 software will be used. Continuous parametric data will be expressed as mean and SD. For categoric parametric data results will be presented in means of frequency and percentage. Comparisons between categoric parameters will be done with test x2. Comparisons between the mean values for continuous parameters with normal distribution will be done via unpaired student's test. Comparisons between categoric parameters will be done with Mann Whitney U test. Normal distribution will be checked with Kolmogorov-Smirnov test. Correlation analysis will be done via Pearson Phi coefficient or Spearman Rho. Statistically significant will be differences with p value < 0.05. Evaluation of correlations between selected variables and cardiovascular events and mortality will be via Kaplan Maier curves.

Study limitations Sympathetic tone evaluation is not feasible during the hyper-acute phase of the syndrome. Systolic and diastolic function of left ventricle prior to the event will not always be available for comparison. Patients with severe comorbidities will probably not be enrolled in the study as it will be difficult to perform the necessary testing.

Estimated research outcome The present study estimates to include patients who express apart from the typical - apical form of the syndrome, as described in previous diagnostic criteria (revised Mayo) patients with basal, mid-ventricular and focal distribution of the systolic dysfunction of the left ventricle. It is interesting to investigate whether the currently available data regarding the sympathetic tone and the typical form of the syndrome apply for the atypical forms. As for the MSNA method, the investigators estimate to re-evaluate it as a means for sympathetic tone evaluation in takotsubo patients but also its potential prognostic value for the severity of syndrome on presentation and long-term morbidity. Regarding the MIBG scan, the investigators expect to reevaluate its value as an index of topical innervation integrity in patients who fulfil the new diagnostic criteria. Moreover, to test whether the hypokinetic area is related with impaired innervation during the subacute phase and permanent changes as expressed with fibrosis in CMR one year after the event.

ELIGIBILITY:
Inclusion Criteria:

* age limits
* Subjects able to provide ICF
* Cases fullfilling the InterTAK criteria with CMR to exclude acute myocarditis or myocardial infarction

Exclusion Criteria:

* age limits
* eGFR < 30ml/min
* Cases diagnosed with acute myocarditis or acute myocardial infarction
* Severe valvular disease not related to TakoTsubo syndrome
* Pacemaker dependent patients
* Contraindications for CMR performance
* Permanent atrial fibrillation
* Neurological conditions related with autonomic failure
* Pregnancy, lactation
* Iodine allergy
* Chronic heart failure with LVEF < 35%
* Any condition related with reduced life expectancy at recruitement
* Cancer on active treatment

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is a prospective, non-interventional observational study which will enroll patients 18-85-year-old, who fulfil the InterTAK diagnostic criteria. The diagnosis will be confirmed with CMR and ECHO which will show the LV systolic recovery. Signed consent form will be obtained and cases that the symptoms were attributed to myocarditis or subendocardial infarction will be excluded. Patients with severe chronic kidney disease (eGFR < 30 ml/min), severe valvular disease, contraindication to perform any of the aforementioned measurements, chronic atrial fibrillation, permanent pacing, autonomic failure, pregnant or breastfeeding women, psychiatric disease which does not allow adequate co-operation or patients with life expectancy less than a year will not be enrolled. The enrolled cases will be followed up for one year. Data will be collected in a specific form (CRF). These include demographic and somatometric data, past medical history, hemodynamics and sympathetic tone measurements.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-10-07 (Estimated); Study Completion 2023-10-07 (Estimated)

PRIMARY OUTCOMES:
Degree of systolic dysfunction at baseline regarding the sympathetic tone activity | 14 days (subacute phase)
  Assesses the impact of sympathetic tone activity over the subacute phase of syndrome with regards to the degree of the systolic dysfunction during the acute event.
Degree of systolic dysfunction at baseline with regards to the sympathetic tone activity 12 months after the event | 12 months after the acute event
  Assesses the impact of sympathetic tone activity over the subacute phase of syndrome as well as one year after the acute episode with regards to the degree of the systolic dysfunction during the acute event.

SECONDARY OUTCOMES:
Degree of diastolic dysfunction at 12 months regarding the sympathetic tone activity at baseline | 12 months follow up
  Assesses the impact of sympathetic tone activity during the subacute phase of syndrome on the diastolic function one year after the acute episode using ECHO features, as well as retrospective echo data from the patient's history regarding diastolic function prior to the event.
Degree of diastolic dysfunction at 12 months regarding the sympathetic tone activity at baseline | 12 months follow up
  Assesses the impact of sympathetic tone activity during the subacute phase of syndrome on the diastolic function one year after the acute episode using CMR features, as well as retrospective echo data from the patient's history regarding diastolic function prior to the event.
Degree of diastolic dysfunction at 12 months regarding the change of sympathetic tone activity during the follow up period | 12 months follow up
  Assesses the impact of sympathetic tone activity change during follow up on the diastolic function one year after the acute episode using ECHO features, as well as retrospective echo data from the patient's history regarding diastolic function prior to the event.
Degree of diastolic dysfunction at 12 months regarding the change of sympathetic tone activity during the follow up period | 12 months follow up
  Assesses the impact of sympathetic tone activity change during follow up on the diastolic function one year after the acute episode using CMR features, as well as retrospective echo data from the patient's history regarding diastolic function prior to the event.
Degree of myocardial fibrosis at 12 months regarding the sympathetic tone activity at baseline | 12 months follow up
  Assesses the impact of sympathetic tone activity over the subacute phase of syndrome with regards to the degree of fibrosis found on CMR one year after the acute episode, if any.
Degree of myocardial fibrosis at 12 months regarding the change of sympathetic tone activity during the follow up period | 12 months follow up
  Assesses the impact of sympathetic tone activity change over the follow up period with regards to the degree of fibrosis found on CMR one year after the acute episode, if any.
Degree of cardiac innervation defect regarding the sympathetic tone activity at baseline | 14 days (subacute phase)
  In the subgroup of patients who will undergo MIBG scan, it assesses the impact of sympathetic tone activity on the cardiac innervation defect derived by the MIBG scan.
Cardiac innervation defect at baseline regarding the diastolic function at 12 months | 12 months follow up
  In the subgroup of patients who will undergo MIBG scan, it assesses the impact of the cardiac innervation defect derived by the MIBG scan during the subacute phase, on the degree of diastolic dysfunction one year after the acute event.
Remaining cardiac innervation defect at baseline regarding the degree of myocardial fibrosis at 12 months | 12 months follow up
  In the subgroup of patients who will undergo MIBG scan, it assesses the impact of the cardiac innervation defect derived by the MIBG scan during the subacute phase, on the degree of myocardial fibrosis one year after the acute event.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos P Tsioufis, Professor, Principal Investigator — 1st Cardiolgogy Clinic, Hippocratio General Hospital of Athens, National and Kapodistrian University of Athens, Greece
Locations (1):
- First Cardiology Clinic, Hippocration General Hospital, National and Kapodistrian University of Athens, Athens, Greece, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Anonymised data may be available for research purposes under the GDPR regulations.

REFERENCES:
- [Background] Y-Hassan S. Acute cardiac sympathetic disruption in the pathogenesis of the takotsubo syndrome: a systematic review of the literature to date. Cardiovasc Revasc Med. 2014 Jan;15(1):35-42. doi: 10.1016/j.carrev.2013.09.008. Epub 2013 Oct 18. PMID 24140050
- [Background] Pollick C, Cujec B, Parker S, Tator C. Left ventricular wall motion abnormalities in subarachnoid hemorrhage: an echocardiographic study. J Am Coll Cardiol. 1988 Sep;12(3):600-5. doi: 10.1016/s0735-1097(88)80044-5. PMID 3403818
- [Background] Pavlovitch JH, Rizk-Rabin M, Jaffray P, Hoehn H, Poot M. Characteristics of homogeneously small keratinocytes from newborn rat skin: possible epidermal stem cells. Am J Physiol. 1991 Dec;261(6 Pt 1):C964-72. doi: 10.1152/ajpcell.1991.261.6.C964. PMID 1767823
- [Background] Wittstein IS, Thiemann DR, Lima JA, Baughman KL, Schulman SP, Gerstenblith G, Wu KC, Rade JJ, Bivalacqua TJ, Champion HC. Neurohumoral features of myocardial stunning due to sudden emotional stress. N Engl J Med. 2005 Feb 10;352(6):539-48. doi: 10.1056/NEJMoa043046. PMID 15703419
- [Background] Ghadri JR, Wittstein IS, Prasad A, Sharkey S, Dote K, Akashi YJ, Cammann VL, Crea F, Galiuto L, Desmet W, Yoshida T, Manfredini R, Eitel I, Kosuge M, Nef HM, Deshmukh A, Lerman A, Bossone E, Citro R, Ueyama T, Corrado D, Kurisu S, Ruschitzka F, Winchester D, Lyon AR, Omerovic E, Bax JJ, Meimoun P, Tarantini G, Rihal C, Y-Hassan S, Migliore F, Horowitz JD, Shimokawa H, Luscher TF, Templin C. International Expert Consensus Document on Takotsubo Syndrome (Part II): Diagnostic Workup, Outcome, and Management. Eur Heart J. 2018 Jun 7;39(22):2047-2062. doi: 10.1093/eurheartj/ehy077. PMID 29850820
- [Background] Ghadri JR, Wittstein IS, Prasad A, Sharkey S, Dote K, Akashi YJ, Cammann VL, Crea F, Galiuto L, Desmet W, Yoshida T, Manfredini R, Eitel I, Kosuge M, Nef HM, Deshmukh A, Lerman A, Bossone E, Citro R, Ueyama T, Corrado D, Kurisu S, Ruschitzka F, Winchester D, Lyon AR, Omerovic E, Bax JJ, Meimoun P, Tarantini G, Rihal C, Y-Hassan S, Migliore F, Horowitz JD, Shimokawa H, Luscher TF, Templin C. International Expert Consensus Document on Takotsubo Syndrome (Part I): Clinical Characteristics, Diagnostic Criteria, and Pathophysiology. Eur Heart J. 2018 Jun 7;39(22):2032-2046. doi: 10.1093/eurheartj/ehy076. PMID 29850871
- [Background] Sharkey SW, Maron BJ. Epidemiology and clinical profile of Takotsubo cardiomyopathy. Circ J. 2014;78(9):2119-28. doi: 10.1253/circj.cj-14-0770. Epub 2014 Aug 5. PMID 25099475
- [Background] Templin C, Ghadri JR, Diekmann J, Napp LC, Bataiosu DR, Jaguszewski M, Cammann VL, Sarcon A, Geyer V, Neumann CA, Seifert B, Hellermann J, Schwyzer M, Eisenhardt K, Jenewein J, Franke J, Katus HA, Burgdorf C, Schunkert H, Moeller C, Thiele H, Bauersachs J, Tschope C, Schultheiss HP, Laney CA, Rajan L, Michels G, Pfister R, Ukena C, Bohm M, Erbel R, Cuneo A, Kuck KH, Jacobshagen C, Hasenfuss G, Karakas M, Koenig W, Rottbauer W, Said SM, Braun-Dullaeus RC, Cuculi F, Banning A, Fischer TA, Vasankari T, Airaksinen KE, Fijalkowski M, Rynkiewicz A, Pawlak M, Opolski G, Dworakowski R, MacCarthy P, Kaiser C, Osswald S, Galiuto L, Crea F, Dichtl W, Franz WM, Empen K, Felix SB, Delmas C, Lairez O, Erne P, Bax JJ, Ford I, Ruschitzka F, Prasad A, Luscher TF. Clinical Features and Outcomes of Takotsubo (Stress) Cardiomyopathy. N Engl J Med. 2015 Sep 3;373(10):929-38. doi: 10.1056/NEJMoa1406761. PMID 26332547
- [Background] Stiermaier T, Thiele H, Eitel I. Long-term excess mortality in Takotsubo syndrome: is it justified to charge Takotsubo for the excess long-term mortality?: Reply. Eur J Heart Fail. 2016 Jul;18(7):879. doi: 10.1002/ejhf.573. Epub 2016 May 30. No abstract available. PMID 27241281
- [Background] Scally C, Rudd A, Mezincescu A, Wilson H, Srivanasan J, Horgan G, Broadhurst P, Newby DE, Henning A, Dawson DK. Persistent Long-Term Structural, Functional, and Metabolic Changes After Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2018 Mar 6;137(10):1039-1048. doi: 10.1161/CIRCULATIONAHA.117.031841. Epub 2017 Nov 11. PMID 29128863
- [Background] Nowak R, Fijalkowska M, Gilis-Malinowska N, Jaguszewski M, Galaska R, Rojek A, Narkiewicz K, Gruchala M, Fijalkowski M. Left ventricular function after takotsubo is not fully recovered in long-term follow-up: A speckle tracking echocardiography study. Cardiol J. 2017;24(1):57-64. doi: 10.5603/CJ.a2017.0001. Epub 2017 Jan 10. PMID 28070881
- [Background] Bratis K. Cardiac Magnetic Resonance in Takotsubo Syndrome. Eur Cardiol. 2017 Aug;12(1):58-62. doi: 10.15420/ecr.2017:7:2. PMID 30416553
- [Background] Nakajima K, Scholte AJHA, Nakata T, Dimitriu-Leen AC, Chikamori T, Vitola JV, Yoshinaga K. Cardiac sympathetic nervous system imaging with 123I-meta-iodobenzylguanidine: Perspectives from Japan and Europe. J Nucl Cardiol. 2017 Jun;24(3):952-960. doi: 10.1007/s12350-017-0818-y. Epub 2017 Mar 13. PMID 28290098
- [Background] Pina IL, Carson P, Lindenfeld J, Archambault WT, Jacobson AF. Persistence of 123I-mIBG Prognostic Capability in Relation to Medical Therapy in Heart Failure (from the ADMIRE-HF Trial). Am J Cardiol. 2017 Feb 1;119(3):434-439. doi: 10.1016/j.amjcard.2016.10.024. Epub 2016 Oct 31. PMID 27912890
- [Background] Akashi YJ, Nakazawa K, Sakakibara M, Miyake F, Musha H, Sasaka K. 123I-MIBG myocardial scintigraphy in patients with "takotsubo" cardiomyopathy. J Nucl Med. 2004 Jul;45(7):1121-7. PMID 15235057
- [Background] Burgdorf C, von Hof K, Schunkert H, Kurowski V. Regional alterations in myocardial sympathetic innervation in patients with transient left-ventricular apical ballooning (Tako-Tsubo cardiomyopathy). J Nucl Cardiol. 2008 Jan-Feb;15(1):65-72. doi: 10.1016/j.nuclcard.2007.08.005. Epub 2007 Oct 29. PMID 18242481
- [Background] Christensen TE, Bang LE, Holmvang L, Skovgaard DC, Oturai DB, Soholm H, Thomsen JH, Andersson HB, Ghotbi AA, Ihlemann N, Kjaer A, Hasbak P. (123)I-MIBG Scintigraphy in the Subacute State of Takotsubo Cardiomyopathy. JACC Cardiovasc Imaging. 2016 Aug;9(8):982-90. doi: 10.1016/j.jcmg.2016.01.028. Epub 2016 Jun 22. PMID 27344416
- [Background] Sverrisdottir YB, Schultz T, Omerovic E, Elam M. Sympathetic nerve activity in stress-induced cardiomyopathy. Clin Auton Res. 2012 Dec;22(6):259-64. doi: 10.1007/s10286-012-0162-x. Epub 2012 Apr 11. PMID 22492095
- [Background] Vaccaro A, Despas F, Delmas C, Lairez O, Lambert E, Lambert G, Labrunee M, Guiraud T, Esler M, Galinier M, Senard JM, Pathak A. Direct evidences for sympathetic hyperactivity and baroreflex impairment in Tako Tsubo cardiopathy. PLoS One. 2014 Mar 25;9(3):e93278. doi: 10.1371/journal.pone.0093278. eCollection 2014. PMID 24667435